CLINICAL TRIAL: NCT00296335
Title: A Phase III Randomized Controlled Trial of Adjuvant Chemotherapy for Advanced Gastric Adenocarcinoma
Brief Title: Trial of Adjuvant Chemotherapy for Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Ulsan University Hospital (Other); Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC-ONCGI-0204
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Stomach Cancer
Keywords: Stomach cancer; Adjuvant chemotherapy; Mitomycin; Cisplatin; Doxifluridine
MeSH Terms: conditions — Stomach Neoplasms | interventions — Mitomycin; doxifluridine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitomycin and doxifluridine (Active Comparator): Mitomycin-C 20mg/m2 intravenously (day 1), Doxifluridine 460-600mg/m2/day per oral (day 28-day 84)
  Interventions: Drug: Mitomycin and doxifluridine
- Mitomycin, doxifluridine and cisplatin (Experimental): Mitomycin-C 20mg/m2 intravenously (day 1), Doxifluridine 460-600mg/m2/day per oral (day 28- day 336), Cisplatin 60mg/m2 intravenously (day 28, day 56, day 84, day 112, day 140, and day 168)
  Interventions: Drug: Mitomycin, doxifluridine and cisplatin

INTERVENTIONS:
Drug: Mitomycin, doxifluridine and cisplatin — Mitomycin-C 20mg/m2 intravenously (day 1), Doxifluridine 460-600mg/m2/day per oral (day 28- day 336), Cisplatin 60mg/m2 intravenously (day 28, day 56, day 84, day 112, day 140, and day 168)
  Arms: Mitomycin, doxifluridine and cisplatin
Drug: Mitomycin and doxifluridine — Mitomycin-C 20mg/m2 intravenously (day 1), Doxifluridine 460-600mg/m2/day per oral (day 28-day 84)
  Arms: Mitomycin and doxifluridine

SUMMARY:
This is a phase III randomized study designed to evaluate the efficacy of mitomycin, doxifluridine, and cisplatin compared to mitomycin and doxifluridine.

DETAILED DESCRIPTION:
Stomach cancer is the most common cancer in Korea and one of the major health problems worldwide. The most effective treatment for gastric cancer is curative surgical resection of primary tumor. However, a substantial number of patients eventually die of recurrences after curative resection. A number of randomized trials investigating the role of adjuvant chemotherapy have been conducted. However, the efficacy of adjuvant chemotherapy is still controversial and varied between Western and Asian trials. Meta-analysis of Western trials didn't demonstrate the benefit of adjuvant chemotherapy after curative resection. Conversely, some Asian studies have demonstrated the efficacy of adjuvant chemotherapy after curative resection. In a previous study, mitomycin plus tegafur prolonged the survival in resected gastric cancer compared to no treatment.

This study is designed to evaluate the efficacy of mitomycin, cisplatin and prolonged treatment with doxifluridine compared to mitomycin plus doxifluridine.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven gastric adenocarcinoma
* Curative resection was done
* stage II, IIIA, IIIB, IV (including T4, lesions or N3, but excluding M1 lymph node metastasis)
* age: 18-69 years old
* Performance status: ECOG 0-2
* Adequate bone marrow function (WBC ≥ 4,000/ul, platelet count ≥ 100,000/ul, hemoglobin ≥ 10 g/dl)
* Adequate renal function (serum creatinine≤ 1.5)
* Adequate liver function (serum bilirubin ≤1.5 mg/dl, AST/ALT ≤ 3 x normal upper limit)
* Written informed consent was signed by the patient

Exclusion Criteria:

* Previous chemotherapy or radiotherapy
* Active ongoing infection which antibiotic treatment is needed
* Pregnant or lactating women
* Psychosis or convulsion disorder
* Ascites in preoperative abdomen CT
* Systemic disease which interfere the administration of chemotherapy
* Previous history of other malignancy except cured non-malignant skin cancer and uterine cervical cancer in situ

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Actual)
Dates: Start 2002-02; Primary Completion 2007-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, M.D.,Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: AMC0201 was an open-label, prospective randomised phase 3 clinical trial conducted at three centres (Asan medical center, Hallym University medical center, and Ulsan university hospital) in Korea. Patients were enrolled between February 2002 and August 2006
Pre-assignment Details: All enrolled patients received study treatments
Period: Overall Study
Arm/Group | Mitomycin and Doxifluridine | Mitomycin, Doxifluridine and Cisplatin
Started | 424 | 431
Completed | 394 | 309
Not Completed | 30 | 122
Not completed — Recurrence | 3 | 51
Not completed — Adverse Event | 17 | 27
Not completed — Lost to Follow-up | 7 | 33
Not completed — Physician Decision | 3 | 11

BASELINE CHARACTERISTICS:
Population: All enrolled patients were included in the analysis.
Groups:
- Mitomycin and Doxifluridine: Mitomycin-C 20mg/m2 intravenously (day 1), Doxifluridine 460-600mg/m2/day per oral (day 28- day 336), Cisplatin 60mg/m2 intravenously (day 28, day 56, day 84, day 112, day 140, and day 168)
- Mitomycin, Doxifluridine and Cisplatin: Experimental armMitomycin-C 20mg/m2 intravenously (day 1), Doxifluridine 460-600mg/m2/day per oral (day 28- day 336), Cisplatin 60mg/m2 intravenously (day 28, day 56, day 84, day 112, day 140, and day 168)
- Total: Total of all reporting groups
Arm/Group | Mitomycin and Doxifluridine | Mitomycin, Doxifluridine and Cisplatin | Total
Number analyzed (Participants) | 424 | 431 | 855
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 361 | 380 | 741
  >=65 years | 63 | 51 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.6) | 53.3 (10.1) | 53.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 137 | 267
  Male | 294 | 294 | 588
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 424 | 431 | 855

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival Rate
Description: Relapse-free survival at 3 years was defined as the proportion of patients who did not show an evidence of disease recurrence after 3 years of surgery.
  Relapse was defined as any new tumor lesion.
Time Frame: 3 years
Population: Intention-to treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Mitomycin Plus Short-term Fluoropyrimidine: Mitomycin-C 20mg/m2 intravenously (day 1), Doxifluridine 460-600mg/m2/day per oral (day 28-day 84)
- Mitomycin Plus Long-term Fluoropyrimidine and Monthly Cisplati: Mitomycin-C 20mg/m2 intravenously (day 1), Doxifluridine 460-600mg/m2/day per oral (day 28- day 336), Cisplatin 60mg/m2 intravenously (day 28, day 56, day 84, day 112, day 140, and day 168)
Arm/Group | Mitomycin Plus Short-term Fluoropyrimidine | Mitomycin Plus Long-term Fluoropyrimidine and Monthly Cisplati
Number analyzed (Participants) | 424 | 431
percentage of participants | 67.0 [62.5 to 71.5] | 64.9 [60.4 to 69.4]

2. Secondary Outcome: Overall Survival Rate
Description: Overall survival rate at 3 years was defined as the proportion of patients who were alive at 3 years after surgery.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Mitomycin Plus Short-term Fluoropyrimidine: Control arm
- Mitomycin Plus Long-term Fluoropyrimidine and Monthly Cisplati: Experimental arm
Arm/Group | Mitomycin Plus Short-term Fluoropyrimidine | Mitomycin Plus Long-term Fluoropyrimidine and Monthly Cisplati
Number analyzed (Participants) | 424 | 431
percentage of participants | 76.9 [72.9 to 80.9] | 73.1 [68.9 to 77.3]

3. Secondary Outcome: Number of Patients With Adverse Events
Description: Per National Cancer Institute Common Toxicity Criteria version 2.0, up to 3 years
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | Mitomycin Plus Short-term Fluoropyrimidine | Mitomycin Plus Long-term Fluoropyrimidine and Monthly Cisplati
Number analyzed (Participants) | 422 | 425
participants
  Neutropenia | 262 | 387
  Anemia | 393 | 413
  Thrombocytopenia | 101 | 156
  Fatigue | 343 | 391
  Diarrhea | 219 | 288
  Nausea | 293 | 371
  Vomiting | 104 | 160

ADVERSE EVENTS:
Arm/Group | Mitomycin Plus Short-term Fluoropyrimidine | Mitomycin Plus Long-term Fluoropyrimidine and Monthly Cisplati
Serious Adverse Events (participants affected / at risk) | 3/422 | 5/425
Other Adverse Events (participants affected / at risk) | 393/422 | 413/425
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitomycin Plus Short-term Fluoropyrimidine (N=422) | Mitomycin Plus Long-term Fluoropyrimidine and Monthly Cisplati (N=425)
Diarrhea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mitomycin Plus Short-term Fluoropyrimidine (N=422) | Mitomycin Plus Long-term Fluoropyrimidine and Monthly Cisplati (N=425)
Neutropenia (Blood and lymphatic system disorders) | 262 | 387
Anemia (Blood and lymphatic system disorders) | 393 | 413
Thrombocytopenia (Blood and lymphatic system disorders) | 101 | 156
Hyperbilirubinemia (Hepatobiliary disorders) | 114 | 162
Fatigue (General disorders) | 343 | 391
Anorexia (General disorders) | 326 | 389
Nausea (Gastrointestinal disorders) | 293 | 371
Vomiting (Gastrointestinal disorders) | 104 | 160
Stomatitis (Gastrointestinal disorders) | 77 | 151
Diarrhea (Gastrointestinal disorders) | 219 | 288
Alopecia (Skin and subcutaneous tissue disorders) | 261 | 334
Neuropathy (Nervous system disorders) | 149 | 301
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 35 | 73
Myalgia (Musculoskeletal and connective tissue disorders) | 109 | 167
Edema (Musculoskeletal and connective tissue disorders) | 44 | 108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No